CLINICAL TRIAL: NCT00208949
Title: A Randomized Comparison of Dendritic Cell Content and T-Cell Phenotype Between G-CSF(Granulocyte Colony-Stimulating Factor)or G-CSF+GM-CSF (Granulocyte Macrophage Colony-Stimulating Factor) for the Mobilization of Normal Allogeneic Peripheral Blood Stem Cell Donors
Brief Title: A Comparison of Dendritic Cell Content and T-Cell Phenotype Between Granulocyte Colony-Stimulating Factor (G-CSF) or G-CSF + Granulocyte Macrophage (GM)-CSF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sagar Lonial, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0693-2002
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-08

CONDITIONS: Hematologic Diseases
Keywords: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Granulocyte Colony-Stimulating Factor; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF(Granulocyte Colony-Stimulating Factor ) (Active Comparator): Single use of G-CSF(Granulocyte Colony-Stimulating Factor ) G-CSF 7.5 µg/kg twice a day
  Interventions: Drug: G-CSF
- Granulocyte CSF+Granulocyte Macrophage CSF (Active Comparator): Combined use of G-CSF(Granulocyte Colony-Stimulating Factor ) and GM-CSF (Granulocyte Macrophage Colony Stimulating Factor) (G-CSF 7.5 µg/kg / GM-CSF 7.5 µg/kg.)
  Interventions: Drug: G-CSF; Drug: GM-CSF

INTERVENTIONS:
Drug: G-CSF — G-CSF, solution given subcutaneously twice per day, total dosage varies by weight.
  Other Names: Rhu
Drug: GM-CSF — GM-CSF, solution given subcutaneously twice per day, total dosage varies by weight.
  Other Names: NSC#617589
  Arms: Granulocyte CSF+Granulocyte Macrophage CSF

SUMMARY:
This is a study involving patients who are undergoing allogeneic peripheral blood stem cell transplantation. Both donors and recipients are being sought for this study.

DETAILED DESCRIPTION:
Patients with leukemia will receive a stem cell transplant, prior to which they will receive medication and/or radiation to destroy all leukemia cells as well as other blood cells. In order to survive this treatment, patients will need to be given the stem cells from another person to replace the blood cells killed by the treatment.

The stem cells given to the recipient will be collected from a relative. To increase the number of stem cells in the relative, he/she is given a growth factor to increase the number of stem cells prior to collection. The standard growth factor used is called G-CSF(Granulocyte Colony-Stimulating Factor ). In this research study, the physician will give the relative either G-CSF or a combination of G-CSF and GM-CSF (Granulocyte Macrophage (GM)) , another type of growth factor. Whether the relative receives G-CSF or GM-CSF will be determined by chance. The donors will be randomized to one or the other. It is not known if the stem cells and white blood cells collected using one or both growth factors results in more cures for this disease and fewer side effects, such as graft-versus-host disease.

The reason for doing the study is to determine if the stem cells and other white blood cells collected are any different when different growth factors are given, and to see how well the patient does. The stem cell transplant will in every other way be the same. The only difference is that if the recipient and donor decide to be in this study, the donor will either be given only G-CSF or the combination of G-CSF and GM-CSF and the recipient will receive the stem cells collected.

ELIGIBILITY:
Inclusion Criteria:

* All normal donors for patients undergoing allogeneic peripheral blood stem cell (PBSC) for hematologic diseases will be invited to participate in this research trial.
* All patients must meet criteria for transplantation.
* Final eligibility will be determined by the health professionals conducting this clinical trial.

Exclusion Criteria:

* Donors for patients undergoing selected or manipulated PBSC grafts are not eligible.
* Donors who are pregnant or lactating females and donors with a known hypersensitivity to either G-CSF or GM-CSF will be excluded from this study.
* Final eligibility will be determined by the health professionals conducting this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-09; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Lonial, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- G-CSF (Granulocyte Colony- Stimulating Factor): Single use of G-CSF
- G-CSF and GM-CSF (Granulocyte Macrophage): Combined use of G-CSF and GM-CSF
Period: Overall Study
Arm/Group | G-CSF (Granulocyte Colony- Stimulating Factor) | G-CSF and GM-CSF (Granulocyte Macrophage)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF (Granulocyte Colony- Stimulating Factor) | G-CSF and GM-CSF (Granulocyte Macrophage) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 2 | 3 | 5
Age, Customized [Median (Full Range); unit: years] | 43 [22 to 64] | 53 [24 to 69] | 49 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 15 | 11 | 26
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Measure the pDC (Plasmacytoid Dendritic Cells )Content of the Graft
Time Frame: at transplant (1 day)
Population: Sample size determinations for this randomized trial were based on a baseline frequency of mDCs(myeloid dendritic cells) and pDCs( plasmacytoid dendritic cells)within the peripheral blood of 0.5% with a SD equal to the mean (0.5%).
Measure: Median (Standard Error); unit: x10 ^ 6 cells/kg
Groups:
- G-CSF (Granulocyte Colony- Stimulating Factor): Single use of G-CSF(Granulocyte Colony-Stimulating Factor ) G-CSF 7.5 µg/kg twice a day
- G-CSF and GM-CSF (Granulocyte Macrophage): Combined use of G-CSF(Granulocyte Colony-Stimulating Factor ) and GM-CSF (Granulocyte Macrophage Colony Stimulating Factor) (G-CSF 7.5 µg/kg / GM-CSF 7.5 µg/kg.)
Arm/Group | G-CSF (Granulocyte Colony- Stimulating Factor) | G-CSF and GM-CSF (Granulocyte Macrophage)
Number analyzed (Participants) | 25 | 25
x10 ^ 6 cells/kg | 4 (1) | 2.5 (1)

2. Secondary Outcome: Median Survival of Recipients of Grafts Mobilized With GM+G+CSF (Granulocyte Colony-Stimulating Factor (G-CSF)+ Granulocyte Macrophage (GM)-CSF) and G-CSF (Granulocyte Colony-Stimulating Factor )at the Time of Last Follow up.
Description: Median overall survival
Time Frame: 5 years
Measure: Median (Full Range); unit: months
Arm/Group | G-CSF (Granulocyte Colony- Stimulating Factor) | G-CSF and GM-CSF (Granulocyte Macrophage)
Number analyzed (Participants) | 25 | 25
months | 38.3 [0 to 60] | 7.3 [0 to 60]

ADVERSE EVENTS:
Arm/Group | G-CSF (Granulocyte Colony- Stimulating Factor) | G-CSF and GM-CSF (Granulocyte Macrophage)
Serious Adverse Events (participants affected / at risk) | 7/25 | 7/25
Other Adverse Events (participants affected / at risk) | 17/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF (Granulocyte Colony- Stimulating Factor) (N=25) | G-CSF and GM-CSF (Granulocyte Macrophage) (N=25)
Death (Blood and lymphatic system disorders) | 7 | 7 — Patients with Leukemia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF (Granulocyte Colony- Stimulating Factor) (N=25) | G-CSF and GM-CSF (Granulocyte Macrophage) (N=25)
Fever (General disorders) | 2 | 9
Bone Pain (Musculoskeletal and connective tissue disorders) | 12 | 19
Injection site redness (Skin and subcutaneous tissue disorders) | 1 | 3
Injected site pain (Musculoskeletal and connective tissue disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes